CLINICAL TRIAL: NCT02612259
Title: A Phase II, Randomized, Double-blind, Placebo-controlled, in Parallel Groups Clinical Trial to Assess the Safety and Efficacy of Dietary Supplementation With Tryptophan to Achieve Weight Loss, and Its Neuropsychological Effects in Adolescent Patients Age 12 to 17 Years With Obesity
Brief Title: A Phase II, Randomized, Double-blind, Placebo-controlled, in Parallel Groups Clinical Trial to Assess the Safety and Efficacy of Dietary Supplementation With Tryptophan to Achieve Weight Loss, and Its Neuropsychological Effects in Adolescents With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSJD-OB-TRP; 2009-016921-32 (EudraCT Number)
Record Dates: First submitted 2015-11-17; First posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Tryptophan; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRYPTOPHAN (Experimental): tryptophan 3.5 mg / kg / day divided in 2 doses, one before breakfast and another one before dinner. Oral administration.
  Total treatment duration for each patient is 6 months.
  Interventions: Dietary Supplement: TRYPTOPHAN
- PLACEBO (Placebo Comparator): lactose capsules 3.5 mg / kg / day divided in 2 doses, one before breakfast and another one before dinner. Oral administration.
  Total treatment duration for each patient is 6 months.
  Interventions: Other: PLACEBO

INTERVENTIONS:
Dietary Supplement: TRYPTOPHAN — at the dose of 3,5 m/kg/ day divided in two capsules
  Arms: TRYPTOPHAN
Other: PLACEBO — at the dose of 3,5 m/kg/ day divided in two capsules
  Other Names: lactose capsules
  Arms: PLACEBO

SUMMARY:
A phase II, randomized, double-blind, placebo-controlled, in parallel groups clinical trial to assess the safety and efficacy of dietary supplementation with tryptophan to achieve weight loss, and its neuropsychological effects in adolescents with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients, attending the Pediatric Endocrinology Service on an out-patient basis.
2. Age from 12 to 17 years, inclusively.
3. Presence of a BMI > or = to 2SD and < or = to 4SD (standard deviations) for their age and sex (Spanish cross-sectional growth reference tables of 2008)
4. Patients must have an educational level that permits adequate communication and must agree to cooperate in all the tests and examinations included in the protocol.
5. Subjects of reproductive potential must use an effective birth control method during the study. Women of reproductive age will be recruited after a negative pregnancy test.
6. The informed consent of the parents or legal representative and of the young adults is required.

Exclusion Criteria:

1. Obesity secondary to an endocrine disease (hypothyroidism, Cushing?s syndrome, polycystic ovary, hypothalamic syndromes, hypogonadism) or the use of medications such as cortisol.
2. Concomitant administration of other psychotrophic medication such as antidepressants or anxiolytics.
3. Patients included in the study must not be taking any vitamins or nutritional supplements or any anti-obesity preparations, including herbal remedies, pharmacy products or homeopathic products.
4. Patients with a known psychiatric disorder.
5. Patients treated with any kind of structured psychotherapy regime.
6. Patients with type 2 DM, arterial hypertension (blood pressure above the 95 percentile for gender and height) or steatotic liver (hypertransaminasemia with echographic image of fatty liver).
7. Patients with any severe food intolerance, or with a known allergy to any of the substances used in the study.
8. Patients in treatment with oral hypoglycemiants.
9. Pregnant or breast-feeding.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in weight by comparing the two groups | From baseline up to 6 months
  to achieve weight loss using Linear Models for Multivariate Outcomes considering as a variables the number of visits, the gender and the group of each patient
Change in systolic and diastolic blood pressure | From baseline up to 6 months
  to achieve improvement of clinical parameters after 6 months of dietary supplementation with tryptophan and determine the difference between the two groups
Change in Body mass index (BMI) defined as wt/ht2 by comparing the two groups | From baseline up to 6 months
  to achieve weight loss using Linear Models for Multivariate Outcomes considering as a variables the number of visits, the gender and the group of each patient
Change in waist/hip ratio by comparing the two groups | From baseline up to 6 months
  to achieve weight loss using Linear Models for Multivariate Outcomes considering as a variables the number of visits, the gender and the group of each patient
Change in Body Mass Index Z score (zBMI) by comparing the two groups | From baseline up to 6 months
  to achieve weight loss using Linear Models for Multivariate Outcomes considering as a variables the number of visits, the gender and the group of each patient

SECONDARY OUTCOMES:
change in total caloric (Kcal) consumption | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient calories intake were measured during visit 1 and visit 7 and then calories levels were compared with the control group.
Change in calorie consumption measuring weight loss (kcal/Kg/days) | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient calories intake were measured during visit 1 and visit 7 and then calories levels were compared with the control group.
Change in protein consumption | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient protein intake were measured during visit 1 and visit 7 and then proteins levels were compared with the control group.
Total Percent of Calories From Protein | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient protein intake were measured during visit 1 and visit 7 and then proteins levels were compared with the control group.
Total fat consumption | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient fat intake were measured (grams) during visit 1 and visit 7 and then fat levels were compared with the control group.
Total Percent of Calories From Fat | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient calories intake were measured during visit 1 and visit 7 and then calories levels were compared with the control group.
Total carbohydrates consumption | From baseline up to 6 months
  to achieve improvement of metabolic parameters, patient carbohydrates intake were measured (grams of carbohydrates) during visit 1 and visit 7 and then carbohydrates levels were compared with the control group.
the mean of lipids concentration (mg/dl) | From baseline up to 6 months
  to achieve improvement of metabolic parameters, the average amount of TSH were measured during visit 1 and visit 7 and then fat levels were compared with the control group. to achieve improvement of metabolic parameters, the average amount of lipids were measured during visit 1 and visit 7 and then fat levels were compared with the control group. The mean of cholesterol both LDL and HDL were considerate for the evaluation.
the amount of Thyroid-stimulating hormone (TSH) concentration (mU/L) | From baseline up to 6 months
  to evaluate the thyroid profile, the average amount of lipids were measured during visit 1 and visit 7 and then TSH levels were compared with the control group.
the amount of thyroxine T4L concentration (pmol/L) | From baseline up to 6 months
  to evaluate the thyroid profile, the average amount of T4L were measured during visit 1 and visit 7 and then T4L levels were compared with the control group.
the amount of creatinine levels (mg/dl) | From baseline up to 6 months
  to evaluate the hepatic profile, the average amount of creatinine were measured during visit 1 and visit 7 and then creatinine levels were compared with the control group.
the amount of Alanine Aminotransferase (ALT) levels (mg/dl) | From baseline up to 6 months
  to assess the hepatic functionality, the average amount of ALT were measured during visit 1 and visit 7 and then ALT mean levels were compared with the control group.
the amount of hemoglobin (g/dl) levels | From baseline up to 6 months
  to assess the renal functionality, the average amount of hemoglobin were measured during visit 1 and visit 7 and then hemoglobin mean levels were compared with the control group.
Change in EuroQoL-5 score over 6 months supplement with tryptophan | From baseline up to 6 months
  to achieve improvement in depression and anxiety after tryptophan administration. Evaluation have been made during Visit 1 and vist 7
Change in the Clinical Global Impressions (CGI) Scale score over 6 months supplement with tryptophan | From baseline up to 6 months
  to achieve improvement in depression and anxiety by comparing the tryptophan group with the placebo group
Change in Children's Manifest Anxiety scale (CMAS) score over 6 months supplement with tryptophan | From baseline up to 6 months
  to achieve improvement in depression and anxiety by comparing the tryptophan group with the placebo group
Change in the Eating Attitudes Test (EAT-40) score | From baseline up to 6 months
  the EAT-40 test is a widely used self-report questionnaire 40-item standardized self-report measure for the assessment of symptoms and concerns characteristic of eating disorders
Change in State-Trait Depression Scales score | From baseline up to 6 months
  The State-Trait Personality Inventory (STPI) is a self-administered questionnaire, consists of eight 10-item subscales: state and trait anxiety, state and trait anger, state and trait curiosity, and state and trait depression. Results from the tryptophan group were compared with the placebo group
Change in Tryptophan plasma level in obese adolescent after 6 months tryptophan administration | From baseline up to 6 months
  For the safety and tolerance assessment of tryptophan supplementation in obese adolescents
Change in Tryptophan/Large neutral aminoacid (LNNA) ratio in obese adolescent plasma after 6 months of tryptophan administration | From baseline up to 6 months
  For the safety and tolerance assessment of tryptophan supplementation in obese adolescents

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ramón Krauel, PI, Principal Investigator — Hospital Sant Joan de Deu